CLINICAL TRIAL: NCT04895462
Title: Safety and Outcomes of Acute Revascularization Treatment in COVID Patients: an International Comparative Study
Brief Title: Acute Revascularization Treatment in Ischemic Stroke Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Larissa University Hospital (Other); Society of Vascular and Interventional Neurology (Unknown); Hospital de Egas Moniz (Other)
Responsible Party: Principal Investigator, Joao Pedro Marto, João Pedro Marto, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CHUV - Stroke&COVID
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Stroke; Covid19
Keywords: Intravenous thrombolysis; Endovascular treatment; Mechanical thrombectomy
MeSH Terms: conditions — Ischemic Stroke; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ischemic Stroke and COVID-19: Ischemic stroke patients with COVID-19 receiving acute recanalization treatment (intravenous thrombolysis and/or endovascular treatment)
- Control group: Ischemic Stroke without COVID-19: Ischemic stroke patients without COVID-19 receiving acute recanalization treatment (intravenous thrombolysis and/or endovascular treatment)

SUMMARY:
Case-series and cohort studies have shown the feasibility of reperfusion therapies in patients with ischemic stroke and COVID-19, but due to the absence of a contemporary control group of non-COVID-19 patients, small sample size or lack of long-term outcome assessment, concerns regarding safety and efficacy of these treatments remain to be clarified. Taking into account its limitations, some studies documented higher rates of endovascular treatment complications such as clot fragmentation with distal embolization and vessel re-oclusion, to be more difficult to achieve recanalization after endovascular treatment, and higher rates of any intracerebral hemmorhage.

The investigators aim is to assess in a large, multicenter and international cohort, the safety and outcomes of acute reperfusion therapies in patients with ischemic stroke and COVID-19, by comparison with a contemporary control group of patients with ischemic stroke and without COVID-19 from the same centers.

ELIGIBILITY:
1. Inclusion Criteria:

   * Consecutive ischemic stroke patients receiving acute recanalization treatment (intravenous thrombolysis and/or endovascular treatment) up to 24 hours since last time since well, and according to local treatment criteria
   * From 1st of March 2020 (for Chinese Centers from 1st January 2020)
2. Exclusion Criteria:

   * Patients without a PCR- or antigen test within the first 7 days after treatment
   * Patients with nosocomial SARS-CoV-2 infection after receiving acute recanalization treatment - PCR- or antigen test becoming positive more than 7 days after treatment
   * Patients with "Suspect/ probable case of SARS-CoV-2 infection" according to the World Health Organization definition
   * Symptomatic cases of SARS-CoV-2 infection with symptoms resolution more than 7 days before treatment
   * Asymptomatic cases of SARS-CoV-2 infection with treatment performed more than 10 days after first positive test for SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Exposed group - Patients with COVID-19
     * Community-acquired confirmed case of SARS-CoV-2 infection either by a positive PCR- or antigen test, and independently of the presence of identifiable COVID-19 compatible symptoms
     * Patient hospitalized due to COVID-19 and with in-hospital stroke
     * Patients with COVID-19 compatible symptoms before reperfusion treatment and with PCR- or antigen test becoming positive within the first 7 days after treatment
  2. Non-exposed group - Patients without COVID-19 ("controls")
     * Patients without COVID-19 compatible symptoms and with negative PCR- or antigen test within the first 7 days after treatment
Sampling Method: Probability Sample
Enrollment: 15128 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Rate of symptomatic intracranial hemorrhage | 36 hours
  Symptomatic parenchymal hemorrhagic transformation according to the ECASS-2 (European-Australasian Acute Stroke Study - II) definition, and/or subarachnoid hemorrhage with ≥4-point worsening in NIHSS (National Institute of Health Stroke Scale)

SECONDARY OUTCOMES:
Rate of any hemorrhagic transformation | 36 hours
  According to the ECASS-2 (European-Australasian Acute Stroke Study - II) definition
Rate of recanalization after endovascular treatment measured by mTICI (modified treatment in cerebral infarction) | End of procedure
  Only in EVT patients
Rate of successful recanalization after endovascular treatment (defined as final mTICI [modified treatment in cerebral infarction] ≥2b) | End of procedure
  Only in EVT patients
Number of passes during endovascular treatment | End of procedure
  Only in EVT patients
Rate of first pass effect during endovascular treatment | End of procedure
  Only in EVT patients
Rate of procedural complication (Arterial perforation, embolization into a previously non-ischemic territory, and re-occlusion) | End of procedure
  Only in EVT patients
Delta NIHSS (National Institute of Health Stroke Scale) at 24 hours | 24 hours
  Difference between admission NIHSS and NIHSS at 24 hours. NIHSS is a scale used to quantify the severity of neurological deficits after stroke: 0 (no signs) to 42 (very severe stroke)
3-month modified Rankin Scale (mRS) | 3 months
  Functional outcome assessed with mRS at 3-month follow-up. The mRS is an ordinal scale that assigns patients among 7 levels of disability: 0 (no symptom) to 5 (severe disability) and 6 (death)
3-month favorable outcome | 3 months
  Favorable outcome defined as modified Rankin Scale (mRS) ≤2 or equal to pre-stroke mRS
3-month mortality | 3 months
  Mortality assessed at 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: João Pedro Marto, MD, Principal Investigator — Stroke Center, Department of Neurology, Lausanne University Hospital, Lausanne, Switzerland and Deparment of Neurology, Hospital de Egas Moniz, Lisbon, Portugal; George Ntaios, MD, PhD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, School of Health Sciences, University of Thessaly, Larissa, Greece; Davide Strambo, MD, Principal Investigator — Stroke Centre, Neurology Service, Lausanne University Hospital, Lausanne, Switzerland; Patrik Michel, MD, Principal Investigator — Stroke Centre, Neurology Service, Lausanne University Hospital, Lausanne, Switzerland
Locations (1):
- Lausanne University Hospital, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Strambo D, Marto JP, Ntaios G, Nguyen TN, Michel P; Global COVID-19 Stroke Registry. Effect of Asymptomatic and Symptomatic COVID-19 on Acute Ischemic Stroke Revascularization Outcomes. Stroke. 2024 Jan;55(1):78-88. doi: 10.1161/STROKEAHA.123.043899. Epub 2023 Dec 22. PMID 38134260
- [Derived] Marto JP, Strambo D, Ntaios G, Nguyen TN, Herzig R, Czlonkowska A, Demeestere J, Mansour OY, Salerno A, Wegener S, Baumgartner P, Cereda CW, Bianco G, Beyeler M, Arnold M, Carrera E, Machi P, Altersberger V, Bonati L, Gensicke H, Bolognese M, Peters N, Wetzel S, Magrico M, Ramos JN, Sargento-Freitas J, Machado R, Maia C, Machado E, Nunes AP, Ferreira P, Pinho E Melo T, Dias MC, Paula A, Correia MA, Castro P, Azevedo E, Albuquerque L, Alves JN, Ferreira-Pinto J, Meira T, Pereira L, Rodrigues M, Araujo AP, Rodrigues M, Rocha M, Pereira-Fonseca A, Ribeiro L, Varela R, Malheiro S, Cappellari M, Zivelonghi C, Sajeva G, Zini A, Gentile M, Forlivesi S, Migliaccio L, Sessa M, La Gioia S, Pezzini A, Sangalli D, Zedde M, Pascarella R, Ferrarese C, Beretta S, Diamanti S, Schwarz G, Frisullo G, Marcheselli S, Seners P, Sabben C, Escalard S, Piotin M, Maier B, Charbonnier G, Vuillier F, Legris L, Cuisenier P, Vodret FR, Marnat G, Liegey JS, Sibon I, Flottmann F, Broocks G, Gloyer NO, Bohmann FO, Schaefer JH, Nolte C, Audebert HJ, Siebert E, Sykora M, Lang W, Ferrari J, Mayer-Suess L, Knoflach M, Gizewski ER, Stolp J, Stolze LJ, Coutinho JM, Nederkoorn P, van den Wijngaard I, De Meris J, Lemmens R, De Raedt S, Vandervorst F, Rutgers MP, Guilmot A, Dusart A, Bellante F, Calleja-Castano P, Ostos F, Gonzalez-Ortega G, Martin-Jimenez P, Garcia-Madrona S, Cruz-Culebras A, Vera R, Matute MC, Fuentes B, Alonso-de-Lecinana M, Rigual R, Diez-Tejedor E, Perez-Sanchez S, Montaner J, Diaz-Otero F, Perez-de-la-Ossa N, Flores-Pina B, Munoz-Narbona L, Chamorro A, Rodriguez-Vazquez A, Renu A, Ayo-Martin O, Hernandez-Fernandez F, Segura T, Tejada-Meza H, Sagarra-Mur D, Serrano-Ponz M, Hlaing T, See I, Simister R, Werring D, Kristoffersen ES, Nordanstig A, Jood K, Rentzos A, Simunek L, Krajickova D, Krajina A, Mikulik R, Cvikova M, Vinklarek J, Skoloudik D, Roubec M, Hurtikova E, Hruby R, Ostry S, Skoda O, Pernicka M, Jurak L, Eichlova Z, Jira M, Kovar M, Pansky M, Mencl P, Palouskova H, Tomek A, Jansky P, Olserova A, Sramek M, Havlicek R, Maly P, Trakal L, Fiksa J, Slovak M, Karlinski MA, Nowak M, Sienkiewicz-Jarosz H, Bochynska A, Wrona P, Homa T, Sawczynska K, Slowik A, Wlodarczyk E, Wiacek M, Tomaszewska-Lampart I, Sieczkowski B, Bartosik-Psujek H, Bilik M, Bandzarewicz A, Dorobek M, Zielinska-Turek J, Nowakowska-Kotas M, Obara K, Urbanowski P, Budrewicz S, Guzinski M, Switonska M, Rutkowska I, Sobieszak-Skura P, Labuz-Roszak BM, Debiec A, Staszewski J, Stepien A, Zwiernik J, Wasilewski G, Tiu C, Terecoasa EO, Radu RA, Negrila A, Dorobat B, Panea C, Tiu V, Petrescu S, Ozdemir A, Mahmoud M, El-Samahy H, Abdelkhalek H, Al-Hashel J, Ismail II, Salmeen A, Ghoreishi A, Sabetay SI, Gross H, Klein P, Abdalkader M, Jabbour P, El Naamani K, Tjoumakaris S, Abbas R, Mohamed GA, Chebl A, Min J, Hovingh M, Tsai JP, Khan M, Nalleballe K, Onteddu S, Masoud H, Michael M, Kaur N, Maali L, Abraham MG, Khandelwal P, Bach I, Ong M, Babici D, Khawaja AM, Hakemi M, Rajamani K, Cano-Nigenda V, Arauz A, Amaya P, Llanos N, Arango A, Vences MA, Barrientos Guerra JD, Caetano R, Martins RT, Scollo SD, Yalung PM, Nagendra S, Gaikwad A, Seo KD, Georgiopoulos G, Nogueira RG, Michel P; Global COVID-19 Stroke Registry. Safety and Outcome of Revascularization Treatment in Patients With Acute Ischemic Stroke and COVID-19: The Global COVID-19 Stroke Registry. Neurology. 2023 Feb 14;100(7):e739-e750. doi: 10.1212/WNL.0000000000201537. Epub 2022 Nov 9. PMID 36351814